CLINICAL TRIAL: NCT00871741
Title: Feasibility Study of GlaxoSmithKline Biologicals' GSK2202083A Vaccine in Healthy Infants at 3, 5 and 11 Months of Age.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to non-approval of IEC to proposed change in locations. Study discontinuation not due to safety/efficacy reasons related to the vaccine.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111761
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-04

CONDITIONS: Tetanus; Poliomyelitis; Neisseria Meningitidis; Haemophilus Influenzae Type b; Diphtheria; Acellular Pertussis; Hepatitis B
Keywords: Combined vaccine; Primary vaccination
MeSH Terms: conditions — Tetanus; Poliomyelitis; Haemophilus Infections; Diphtheria; Hepatitis B | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (2):
- GSK2202083A GROUP (Experimental): Subjects in this group were to receive three doses of GSK2202083A vaccine at 3, 5 and 11 months of age, as an intramuscular injection in the anterolateral quadrant of the right thigh.
  Interventions: Biological: GSK2202083A vaccine
- INFANRIX + MENJUGATE GROUP (Active Comparator): Subjects in this group were to receive three doses of Infanrix™ hexa vaccine at 3, 5 and 11 months of age, and two doses of Menjugate® vaccine at 3 and 5 months of age, as an intramuscular injection in the anterolateral quadrant of the right thigh.
  Interventions: Biological: Infanrix hexa; Biological: Menjugate

INTERVENTIONS:
Biological: GSK2202083A vaccine — Intramuscular, three doses
  Arms: GSK2202083A GROUP
Biological: Infanrix hexa — Intramuscular, three doses
  Arms: INFANRIX + MENJUGATE GROUP
Biological: Menjugate — Intramuscular, two doses
  Arms: INFANRIX + MENJUGATE GROUP

SUMMARY:
This study will evaluate the safety and immunogenicity of GSK Biologicals' GSK2202083A vaccine given as a three-dose vaccination course at 3, 5 and 11 months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant between, and including, 8 and 16 weeks at the time of the first vaccination.
* Born after a gestation period of 36 to 42 weeks inclusive.
* Subjects who the investigator believes that their parents/ guardians can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to randomisation, or planned administration from randomisation to study Visit 3, or from 30 days before to 30 days after study Visit 4, with the exception of influenza and human rotavirus vaccines. The administration of other vaccines, including conjugated pneumococcal vaccine, is allowed during the period from one day after study Visit 3 to 31 days before study Visit 4.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis, Hib and/or MenC vaccination or disease, including HBV vaccination at birth.
* History of seizures or progressive neurological disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.

The following condition is temporary or self-limiting, and a subject may be vaccinated once the condition has resolved if no other exclusion criteria is met:

• Current febrile illness or axillary temperature >= 38.5 ºC or other moderate to severe illness within 24 hours of study vaccine administration

Ages: 8 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2009-04-01; Primary Completion 2009-06-25 (Actual); Study Completion 2009-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Slovakia (7):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Dolný Kubín
  - GSK Investigational Site, Dunajská Streda
  - GSK Investigational Site, Nové Zámky
  - GSK Investigational Site, Ružomberok
  - GSK Investigational Site, Štúrovo
  - GSK Investigational Site, Trnava

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 111761 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111761 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111761 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111761 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111761 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111761 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111761 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Infanrix + Menjugate Group: Subjects in this group were to receive three doses of Infanrix hexa vaccine at 3, 5 and 11 months of age, and two doses of Menjugate vaccine at 3 and 5 months of age, as an intramuscular injection in the anterolateral quadrant of the right thigh.
Period: Overall Study
Arm/Group | GSK2202083A Group | Infanrix + Menjugate Group
Started | 9 | 7
Completed | 0 | 0
Not Completed | 9 | 7
Not completed — Premature study termination | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2202083A Group | Infanrix + Menjugate Group | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 12.8 (2.28) | 13.9 (1.57) | 13.28 (2.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Anti-PRP Antibody Concentrations ≥ 0.15 mg/mL
Description: As the study was terminated, no blood samples were taken. Hence no immunogenicity analyses were done.
Time Frame: At Month 3
Arm/Group | GSK2202083A Group | Infanrix + Menjugate Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited Local Symptoms
Description: The solicited local symptoms assessed were pain, redness and swelling. Any = any solicited local symptom irrespective of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
  Subjects from Control Group did not receive the second study vaccination dose due to study termination.
Time Frame: During the 8-day (Days 0-7) post-vaccination period following each dose and across doses
Population: The analyses were performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix + Menjugate Group
Number analyzed (Participants) | 9 | 7
Participants
  Any pain, Dose 1 | 2 | 2
  Grade 3 pain, Dose 1 | 0 | 0
  Any redness, Dose 1 | 4 | 4
  Grade 3 redness, Dose 1 | 0 | 0
  Any swelling, Dose 1 | 3 | 1
  Grade 3 swelling, Dose 1 | 1 | 1
  Any pain, Dose 2: number analyzed (Participants) | 1 | 0
  Any pain, Dose 2 | 0 |
  Grade 3 pain, Dose 2: number analyzed (Participants) | 1 | 0
  Grade 3 pain, Dose 2 | 0 |
  Any redness, Dose 2: number analyzed (Participants) | 1 | 0
  Any redness, Dose 2 | 0 |
  Grade 3 redness, Dose 2: number analyzed (Participants) | 1 | 0
  Grade 3 redness, Dose 2 | 0 |
  Any swelling, Dose 2: number analyzed (Participants) | 1 | 0
  Any swelling, Dose 2 | 0 |
  Grade 3 swelling, Dose 2: number analyzed (Participants) | 1 | 0
  Grade 3 swelling, Dose 2 | 0 |
  Any pain, Across doses | 2 | 2
  Grade 3 pain, Across doses | 0 | 0
  Any redness, Across doses | 4 | 4
  Grade 3 redness, Across doses | 0 | 0
  Any swelling, Across doses | 3 | 1
  Grade 3 swelling, Across doses | 1 | 1

3. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: The solicited general symptoms assessed were drowsiness, irritability, loss of appetite and temperature.
  Any = any general symptom irrespective of intensity grade and relationship to vaccination.
  Grade 3 Irritability = crying that could not be comforted/prevented normal activity.
  Grade 3 Drowsiness = drowsiness that prevented normal activity. Grade 3 Loss of Appetite = did not eat at all. Related = symptoms assessed by the investigator as causally related to vaccination.
  Subjects from Control Group did not receive the second study vaccination dose due to study termination.
Time Frame: During the 8-day (Days 0-7) post-vaccination period following each dose and across doses
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix + Menjugate Group
Number analyzed (Participants) | 9 | 7
Participants
  Any drowsiness, Dose 1 | 1 | 1
  Grade 3 drowsiness, Dose 1 | 0 | 0
  Related drowsiness, Dose 1 | 1 | 0
  Any irritability, Dose 1 | 4 | 4
  Grade 3 irritability, Dose 1 | 0 | 0
  Related irritability, Dose 1 | 4 | 3
  Any loss of appetite, Dose 1 | 2 | 1
  Grade 3 loss of appetite, Dose 1 | 0 | 0
  Related loss of appetite, Dose 1 | 2 | 1
  Any temperature, Dose 1 | 4 | 1
  Grade 3 temperature (>39.0°C), Dose 1 | 0 | 0
  Related temperature, Dose 1 | 4 | 1
  Any drowsiness, Dose 2: number analyzed (Participants) | 1 | 0
  Any drowsiness, Dose 2 | 0 |
  Grade 3 drowsiness, Dose 2: number analyzed (Participants) | 1 | 0
  Grade 3 drowsiness, Dose 2 | 0 |
  Related drowsiness, Dose 2: number analyzed (Participants) | 1 | 0
  Related drowsiness, Dose 2 | 0 |
  Any irritability, Dose 2: number analyzed (Participants) | 1 | 0
  Any irritability, Dose 2 | 0 |
  Grade 3 irritability, Dose 2: number analyzed (Participants) | 1 | 0
  Grade 3 irritability, Dose 2 | 0 |
  Related irritability, Dose 2: number analyzed (Participants) | 1 | 0
  Related irritability, Dose 2 | 0 |
  Any loss of appetite, Dose 2: number analyzed (Participants) | 1 | 0
  Any loss of appetite, Dose 2 | 0 |
  Grade 3 loss of appetite, Dose 2: number analyzed (Participants) | 1 | 0
  Grade 3 loss of appetite, Dose 2 | 0 |
  Related loss of appetite, Dose 2: number analyzed (Participants) | 1 | 0
  Related loss of appetite, Dose 2 | 0 |
  Any temperature, Dose 2: number analyzed (Participants) | 1 | 0
  Any temperature, Dose 2 | 1 |
  Grade 3 temperature (>39.0°C), Dose 2: number analyzed (Participants) | 1 | 0
  Grade 3 temperature (>39.0°C), Dose 2 | 0 |
  Related temperature, Dose 2: number analyzed (Participants) | 1 | 0
  Related temperature, Dose 2 | 1 |
  Any drowsiness, Across doses | 1 | 1
  Grade 3 drowsiness, Across doses | 0 | 0
  Related drowsiness, Across doses | 1 | 0
  Any irritability, Across doses | 4 | 4
  Grade 3 irritability, Across doses | 0 | 0
  Related irritability, Across doses | 4 | 3
  Any loss of appetite, Across doses | 2 | 1
  Grade 3 loss of appetite, Across doses | 0 | 0
  Related loss of appetite, Across doses | 2 | 1
  Any temperature, Across doses | 4 | 1
  Grade 3 temperature (>39.0°C), Across doses | 0 | 0
  Related temperature, Across doses | 4 | 1

4. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events AE(s)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix + Menjugate Group
Number analyzed (Participants) | 9 | 7
Participants | 2 | 3

5. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Month 0 to Month 9)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix + Menjugate Group
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 8-day (Days 0-7) post-vaccination period. AEs: during the 31-day (Days 0-30) post-vaccination period. SAEs: Throughout the entire study period (from Month 0 up to Month 9).
Arm/Group | GSK2202083A Group | Infanrix + Menjugate Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 5/9 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2202083A Group (N=9) | Infanrix + Menjugate Group (N=7)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Pain (General disorders) | 2 | 2
Redness (General disorders) | 4 | 4
Swelling (General disorders) | 3 | 1
Drowsiness (General disorders) | 1 | 1
Irritability (General disorders) | 4 | 4
Loss of appetite (General disorders) | 2 | 1
Temperature (General disorders) | 4 | 1
Pyrexia (General disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.